CLINICAL TRIAL: NCT02256098
Title: A Clinical Randomized Controlled RSA Trial Comparing the Cemented ATTUNE™ Fixed Bearing Cruciate Retaining Knee System With the Cemented PFC Sigma Fixed Bearing Cruciate Retaining Knee System
Brief Title: RSA RCT: ATTUNE™ TKA Versus PFC Sigma TKA
Acronym: APKnee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Medical Center Haaglanden (Other); DePuy International (Industry)
Responsible Party: Principal Investigator, R.G.H.H. Nelissen, Prof. PhD MD Head of the Department of Orthopaedics, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P14.142
Record Dates: First submitted 2014-09-23; First posted 2014-10-03 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Osteoarthritis Arthritis; Joint Diseases; Musculoskeletal Diseases; Rheumatic Diseases
Keywords: Comparative Study; Knee Prosthesis; Prosthesis Design; Treatment Outcome; Follow-Up Studies; Arthroplasty, Replacement, Knee/methods
MeSH Terms: conditions — Joint Diseases; Musculoskeletal Diseases; Rheumatic Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ATTUNE™ (Experimental): Total Knee Replacement Surgery with ATTUNE™ Knee Prosthesis by DePuy
  Interventions: Device: ATTUNE™ Knee Prosthesis by DePuy
- PFC Sigma (Active Comparator): Total Knee Replacement Surgery with PFC Sigma Knee Prosthesis by DePuy
  Interventions: Device: PFC Sigma Knee Prosthesis by DePuy

INTERVENTIONS:
Device: ATTUNE™ Knee Prosthesis by DePuy — Total Knee Replacement (TKR) Surgery with ATTUNE™ Knee Prosthesis by DePuy
  Arms: ATTUNE™
Device: PFC Sigma Knee Prosthesis by DePuy — Total Knee Replacement Surgery with PFC Sigma Knee Prosthesis by DePuy
  Arms: PFC Sigma

SUMMARY:
The PFC Sigma Knee by DePuy Synthes is an excellent knee replacement with an excellent clinical track record, good survival rates (98% 10 years survival in patients aged < 55 years)(Keenan et al., 2012) and minimal early migration as measured with RSA (0.5mm MTPM at two years follow-up)(von et al., 2009).

The ATTUNE™ Knee by DePuy Synthes is an advancement in knee replacement options. It is designed to provide better range of motion and address the unstable feeling some patients experience during everyday activities, such as stair descent and bending. To date (March 2013), more than 3,500 patients have received an ATTUNE Knee as part of a limited launch and positive feedback was received regarding patient recovery, stability and motion.

The objective of this study is to accurately assess and compare migration, clinical and radiological outcome and patient reported outcomes of two TKR prostheses: the Cemented ATTUNE™ Fixed Bearing Cruciate Retaining Knee System and the Cemented PFC Sigma Fixed Bearing Cruciate Retaining Knee System, both by DePuy Synthes, Warsaw, Indiana, USA. The primary objective of this study is to compare the magnitude and pattern of migration of the prostheses (Femoral and Tibial component). The secondary objective of this study is to compare clinical and radiological outcome of the prostheses and PROMS. The tertiary objective of this study is to compare clinical and radiological outcome and PROMS of the prostheses with migration data.

This study is designed as a single-blind, randomized trial between the ATTUNE™ Knee System and PFC Sigma Knee System. 32 patients with the ATTUNE™ Knee System and 32 patients with PFC Sigma Knee System will be included in this study.

The study population will consist of patients with symptomatic osteoarthritis of the knee scheduled for TKR surgery at the Department of Orthopaedics, Medisch Centrum Haaglanden, The Hague, The Netherlands. Annually 300 TKA procedures are performed in this department, of which about 90% is Osteo Arthritis (OA) and 10% Rheumatoid Arthritis (RA) and other indications. We anticipate that inclusion can be accomplished within a 1 year period and that the total study duration is 3 years.

Main study parameters/endpoints are:

* Migration of the prosthesis with respect to the host bone measured by means of roentgen stereophotogrammetric analysis (RSA).
* Patient Reported Outcome Measures by means of questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Patient is diagnosed with osteoarthritis or rheumatoid arthritis and requiring primary knee arthroplasty
* All consecutive patients ("usual care") are included to prevent selection bias in the migration analysis.
* Patient is capable of giving informed consent and expressing a willingness to comply with this study

Exclusion Criteria:

* The patient has an a-priori risk for a posterior-stabilized total knee arthroplasty.

  * Insufficiency of the posterior cruciate ligament (PCL)
  * Status after patellectomy
  * In case flexion is less than 90 degrees
  * When it is expected that the tibia cut during surgery will compromise the attachment of the PCL (because of bony defects)
* The patient is unable or unwilling to sign the Informed Consent specific to this study
* The patient does not understand the Dutch or English language good enough to participate
* Patients indicated for revision arthroplasty
* When there are not enough markers visible in the baseline RSA photograph and it will not improve by placing the patient in another position, the patient will be excluded from the study (secondary exclusion criteria).

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2017-11-02 (Actual); Study Completion 2017-11-02 (Actual)

PRIMARY OUTCOMES:
Migration, measured by means of RSA. | 2 Years
  Migration (MTPM in mm) of the prosthesis with respect to the host bone measured by means of roentgen stereophotogrammetric analysis (RSA).

SECONDARY OUTCOMES:
EQ-5D | 2 Years
  General Health: EuroQol 5 Dimensional (EQ-5D) Health Questionnaire measured using patient questionnaire
KOOS | 2 Years
  Knee Function: Knee injury and Osteoarthritis Outcome Score (KOOS) measured using patient questionnaire
VAS pain | 2 Years
  - Pain score after activity and during rest; (Likert scale 0-10)
2 Anchor questions | 2 Years
  Two anchor questions (Likert scale 1-7) about change in functioning and pain since surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Rob G Nelissen, Prof. PhD, MD, Principal Investigator — Dep. Orthopaedics, Leiden University Medical Center; Edward R Valstar, Prof. PhD. MSc, Principal Investigator — Dep. Orthopaedics, Leiden University Medical Center; Peter H den Hollander, MD, Principal Investigator — Dep. Orthopaedics, Medisch Centrum Haaglanden
Locations (2):
- Netherlands (2):
  - Leiden University Medical Center, Leiden
  - Medisch Centrum Haaglanden, The Hague